CLINICAL TRIAL: NCT01705990
Title: A Phase I Double-Blind, Randomized, Placebo-Controlled, Dose-Escalation Trial to Evaluate the Safety and Immunogenicity of a Sendai HIV Vaccine SeV-G(NP) Given Intranasally and Ad35-GRIN Administered Intramuscularly in Prime-Boost Regimens in HIV-Uninfected, Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity Study of SeV-G(NP) HIV Vaccine Administered Intranasally and Ad35-GRIN HIV Vaccine Given Intramuscularly in Prime-Boost Regimens in HIV-Uninfected Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI S001
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; HIV vaccine; HIV prevention
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A: SeV-G(NP) followed by Ad35-GRIN (Experimental): SeV-G(NP) (IN) at 2x10^7 CIU at Month 0 followed by Ad35-GRIN (IM) at 1x10^10 vp at Month 4. (Vaccine/Placebo = 12/4)
  Interventions: Biological: SeV-G(NP) (0.2mL, 2x10^7 CIU); Biological: Ad35-GRIN (0.5mL)
- Group B: SeV-G(NP) followed by Ad35-GRIN (Experimental): SeV-G(NP) (IN) at 2x10^8 CIU at Month 0 followed by Ad35-GRIN (IM) at 1x10^10 vp at Month 4. (Vaccine/Placebo = 12/4)
  Interventions: Biological: SeV-G(NP) (0.2mL, 2x10^8 CIU); Biological: Ad35-GRIN (0.5mL)
- Group C: Ad35-GRIN followed by SeV-G(NP) (Experimental): Ad35-GRIN (IM) at 1x10^10 vp at Month 0 followed by SeV-G(NP) (IN) at 2x10^8 CIU at Month 4. (Vaccine/Placebo = 12/4)
  Interventions: Biological: SeV-G(NP) (0.2mL, 2x10^8 CIU); Biological: Ad35-GRIN (0.5mL)
- Group D: SeV-G(NP) only (Experimental): SeV-G(NP) (IN) at 2x10^8 CIU at Month 0 and 4. (Vaccine/Placebo = 12/4)
  Interventions: Biological: SeV-G(NP) (0.2mL, 2x10^8 CIU)

INTERVENTIONS:
Biological: SeV-G(NP) (0.2mL, 2x10^7 CIU) — Delivered intranasally by drops
  Arms: Group A: SeV-G(NP) followed by Ad35-GRIN
Biological: SeV-G(NP) (0.2mL, 2x10^8 CIU) — Delivered intranasally by drops
  Arms: Group B: SeV-G(NP) followed by Ad35-GRIN; Group C: Ad35-GRIN followed by SeV-G(NP); Group D: SeV-G(NP) only
Biological: Ad35-GRIN (0.5mL) — (1x10^10 vp) Delivered intramuscularly by standard syringe and needle injection
  Arms: Group A: SeV-G(NP) followed by Ad35-GRIN; Group B: SeV-G(NP) followed by Ad35-GRIN; Group C: Ad35-GRIN followed by SeV-G(NP)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of Sendai HIV vaccine SeV-G(NP) given intranasally and Ad35-GRIN administered intramuscularly in prime-boost regimens in HIV-uninfected, healthy adult volunteers.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled, dose-escalation trial assessing the safety, tolerability, and immunogenicity of SeV-G(NP) given intranasally by drops and Ad35-GRIN administered intramuscularly in each of four prime-boost regimens.

Volunteers will be screened up to 42 days before the 1st vaccination and will be followed for 12 months after the last vaccine administration (16 months after the first vaccination). It is anticipated that it will take approximately 6 months to enroll the study. Approximately 64 volunteers (48 vaccine and 16 placebo recipients) will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female adults,
* 18 to 50 years of age (21 to 50 years of age for volunteers in Rwanda),
* who do not report high-risk behaviour for HIV infection,
* who are available for the duration of the trial,
* who are willing to undergo HIV testing,
* use an effective method of contraception, and
* who, in the opinion of the principal investigator or designee, understand the study and who provide written informed consent.

Exclusion Criteria:

* confirmed HIV infection,
* pregnancy and lactation,
* significant acute or chronic disease,
* clinically significant laboratory abnormalities,
* recent vaccination or receipt of a blood product,
* previous receipt of an HIV vaccine, and
* previous severe local or systemic reactions to vaccination or history of severe allergic reactions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 16 months approximately
  To evaluate the safety and tolerability of SeV-G(NP) and Ad35-GRIN administered in four prime-boost regimens.

SECONDARY OUTCOMES:
Shedding | 16 months
  To assess the presence and persistence of the SeV-G(NP) vector and the in vivo genetic integrity of the insert
Immunogenicity | 16 months
  To assess (qualitative and quantitative) immune responses elicited by the different prime-boost regimens.

CONTACTS AND LOCATIONS:
Locations (3):
- Kenya AIDS Vaccine Initiative, Nairobi, Kenya
- Project San Francisco, Kigali, Rwanda
- St. Stephen's Centre, London, United Kingdom

REFERENCES:
- [Derived] Nyombayire J, Anzala O, Gazzard B, Karita E, Bergin P, Hayes P, Kopycinski J, Omosa-Manyonyi G, Jackson A, Bizimana J, Farah B, Sayeed E, Parks CL, Inoue M, Hironaka T, Hara H, Shu T, Matano T, Dally L, Barin B, Park H, Gilmour J, Lombardo A, Excler JL, Fast P, Laufer DS, Cox JH; S001 Study Team. First-in-Human Evaluation of the Safety and Immunogenicity of an Intranasally Administered Replication-Competent Sendai Virus-Vectored HIV Type 1 Gag Vaccine: Induction of Potent T-Cell or Antibody Responses in Prime-Boost Regimens. J Infect Dis. 2017 Jan 1;215(1):95-104. doi: 10.1093/infdis/jiw500. Epub 2016 Oct 17. PMID 28077588
- See also: International AIDS Vaccine Initiative — http://www.iavi.org